CLINICAL TRIAL: NCT00054964
Title: Comparison of Single-dose Efficacy of Albuterol-HFA-BOI and Albuterol-HFA-MDI in Asthmatics With Poor Inhaler Coordinating Ability
Brief Title: Comparative Effectiveness of a Breath-operated Albuterol Inhaler in Asthma Patients With Poor Inhaler Technique
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IXR-202-4-167
Record Dates: First submitted 2003-02-14; First posted 2003-02-17 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol HFA-BOI (Experimental)
  Interventions: Drug: Albuterol HFA-BOI
- Albuterol HFA-MDI (Active Comparator)
  Interventions: Drug: Albuterol HFA-MDI

INTERVENTIONS:
Drug: Albuterol HFA-BOI — Albuterol HFA breath operated inhaler, 90 mcg/sprau
  Arms: Albuterol HFA-BOI
Drug: Albuterol HFA-MDI — Albuterol HFA multi-dose inhaler
  Other Names: Proair HFA-MDI
  Arms: Albuterol HFA-MDI

SUMMARY:
This study was designed to examine the effectiveness of a breath-operated albuterol inhaler in asthma patients who have difficulty using their standard "press-and-breathe" inhaler.

DETAILED DESCRIPTION:
This was a single-center, randomized, open-label, active-controlled, 2-period, 2-sequence, single dose-dose, crossover comparison of the ability of Albuterol BOI-HFA to produce bronchodilation relative to that produced by to albuterol MDI-HFA in at least 12 asthmatics with poor inhaler coordinating ability.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed ≥6 months prior and stable for 4 weeks prior to screening
* Poor inhaler coordination as assessed at screening
* Reversible bronchoconstriction (≥ 12% increase in FEV1)

Exclusion Criteria:

* Albuterol allergy
* Investigational drug within 30 days
* Injected corticosteroid within 6 weeks
* Requires beta-blockers, MAO inhibitors, tricyclic antidepressants, long-acting beta-blockers, steroids other than those inhaled
* Other criterial apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-03-31 (Actual); Primary Completion 2003-08-31 (Actual); Study Completion 2003-08-31 (Actual)

PRIMARY OUTCOMES:
Percent change in SGaw (A measure of the change in specific airway conductance - how hard it is to get air into the lungs) | Pre-dose and +120 minutes

SECONDARY OUTCOMES:
The area-under-the-effect curve of change in SGaw from basline over time | Pre-dose and +120 minutes
The maximum increase in SGaw from baseline over two hours | Baseline through +120 minutes
Time in hours to the maximum increase in SGaw from baseline | Baseline through +120 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Harold Nelson, MD, Principal Investigator — National Jewish Medical Center
Locations (1):
- National Jewish Medical and Research Ceter, Denver, Colorado, United States

REFERENCES:
- [Result] Nelson HS, Wenzel SE, Weisfeld L, Llorens L, Atkinson DC, Stahl EG. Comparison of single-dose efficacy of albuterol-hydrofloroalkane breath-activated inhaler and Nelson HS, Wenzel SE, Weisfeld L, Llorens L, Atkinson DC, Stahl EG. Comparison of single-dose efficacy of albuterol-hydrofloroalkane metered-dose inhaler in asthma patients with poor inhaler coordinating ability. Chest 2008;134:92003S (Abstracts, ACCP Annual Meeting, October 25-30, 2008, Philadelphia, Pennsylvania, USA.